CLINICAL TRIAL: NCT05554718
Title: Evaluation of a Smartphone Application for Self-help for Patients With Social Anxiety Disorder: a Randomized Controlled Study
Brief Title: Evaluation of a Smartphone Application for Self-help for Social Anxiety
Acronym: SMASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goethe University (Other)
Collaborators: Technische Universität Dresden (Other); Mindable Health GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SoPho-App-Evaluation
Record Dates: First submitted 2022-09-12; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Social Anxiety

STUDY DESIGN:
Intervention Model Description: Comparison of self-help app only, self-help app plus accompanying therapy sessions, and waitlist control group
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to the conditions, but blinding of participant and care provider is not possible due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App condition (Experimental): All participants will receive access to the developed social anxiety disorder (SAD) treatment app for 12 weeks.
  Interventions: Behavioral: Self-help Smartphone App
- App with accompanying therapy sessions (Experimental): In addition to being able to use the app to treat social anxiety over a 12-week period, participants will receive a total of 8 video therapy sessions based on cognitive behavioral therapy to accompany their use of the app.
  Interventions: Behavioral: Self-help Smartphone App; Behavioral: Therapist-guided App Use
- Waitlist control condition (No Intervention): Delayed use of the mobile application after 12 weeks.

INTERVENTIONS:
Behavioral: Self-help Smartphone App — The app provides a 12-week adaptation of scientifically proven cognitive behavioral therapy techniques for the treatment of SAD and is intended for use as a mobile intervention. The app includes modules such as learning (e.g., creating a model, learning about the maintaining factors), changing the maintaining factors (e.g., safety behaviors), or behavioral experiments.
  Arms: App condition; App with accompanying therapy sessions
Behavioral: Therapist-guided App Use — In addition to using the app, patients receive a total of 8 video-based therapy sessions over the course of 12 weeks. The sessions include topics such as video feedback and behavioral experiments.
  Arms: App with accompanying therapy sessions

SUMMARY:
The present study examines whether a self-help app can reduce symptoms of social anxiety disorder.

DETAILED DESCRIPTION:
The study will test the effectiveness of a newly developed mobile app in treating patients with social anxiety. Participants will be randomly assigned to one of the following groups: app use only, therapist-guided app use, and a wait-list control group. Over a 12-week period, the study will examine whether mobile app use leads to significant reductions in symptoms associated with social anxiety, as well as improvements in secondary outcomes such as quality of life, depression, or psychological impairment.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Social Anxiety Disorder
* Written informed consent before the start of the study
* Age: 18 to 65 years
* Possession of smartphone
* Familiarity with using smartphone apps

Exclusion Criteria:

* Acute suicidality
* Active substance abuse or dependence
* Severe medical conditions (e.g., chronic cardiovascular disease)
* Severe depression
* Psychotic disorder
* Bipolar disorder
* Borderline personality disorder
* Current psychotherapeutic treatment
* Current psychopharmacological treatment
* No proficient skills in the German language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in SAD-related symptom severity measured by the Liebowitz Social Anxiety Scale | change from baseline (week 0) to week 12 (post) and to week 36 (follow-up)
  The LSAS is a clinician-rated interview designed to measure fear and avoidance in different social situations. The situations are rated on scale from 0 ("not at all" or "never") to 3 (severe" or "most of the time"), with higher scores indicating greater symptoms of social anxiety.

SECONDARY OUTCOMES:
Change in SAD-related symptoms measured by the Social Phobia Inventory (SPIN) | change from baseline to week 12 (post) and to week 36 (follow-up)
  The SPIN is a self-report questionnaire designed to assess the amount of discomfort in different situations during the last week. The scale ranges from 0 ("not at all") to 4 ("extremely"). The total score ranges from 0 to 68, with higher scores indicating more severe symptoms of social anxiety.
Change in the Social Phobic Cognition Questionnaire (SPK) | change from baseline to week 12 (post) and to week 36 (follow-up)
  The SPK lists 22 SAD-related beliefs that are rated on two scales: thought frequency, ranging from 1 ("thought never occurs") to 5 ("thought always occurs") and belief rating, ranging from 0 ("I do not believe this thought") to 100 ("I am completely convinced this thought is true"). Higher scores indicate more SAD-related beliefs.
Pain and Disability Index (PDI) | change from baseline to week 12 (post) and to week 36 (follow-up)
  The PDI measures the amount of impairment and distress caused by the mental illness. It consists of 7 different categories (e.g., "Social Activity") that are rated on a scale fom 0 ("no disability") to 10 ("total disability"). Higher scores indicating higher levels of disability.
Beck Depression Inventory - Fast Screen (BDI-FS) | change from baseline to week 12 (post) and to week 36 (follow-up)
  The BDI-FS assesses symptoms of depression using 7 items on a 4-point scale, with higher scores indicating greater severity.
World Health Organization Quality of Life (WHO-QOL-BREF) | change from baseline to week 12 (post) and to week 36 (follow-up)
  The WHO-QOL-BREF measures the overall quality of life and asks for ratings on varying 5-point-scales for different domains like physical health (e.g., "how satisfied are you with..."). Scores for each domain are transformed to a scale of 0 to 100, with higher overall scores indicating a higher quality of life.
Brief Symptom Inventory - 18-item version (BSI-18) | change from baseline to week 12 (post) and to week 36 (follow-up)
  The BSI measures general psychological distress using 18 items like "feelings of loneliness" on a scale from 0 ("not at all") to 4 ("a lot").
Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) | change from baseline to week 12 (post) and to week 36 (follow-up)
  The ACIPS measures the pleasure a person experiences in a social situation with a total of 17 items. The items are rated on a scale from 1 ("very false for me") to 6 ("very true for me"), with higher total scores indicating higher interpersonal pleasure.
Social Pain Questionnaire-5 (SPQ-5) | baseline measurement only (week 0) before intervention starts
  Sensitivity to rejection in social situations are assessed with the Social Pain Questionnaire (SPQ-5). The questionnaire consists of 5 items rating from 0 ("describes me perfectly") to 4 ("not at all"). Higher total scores indicate higher social pain.
Self-developed question regarding skills in using the Internet | baseline measurement only (week 0) before intervention starts
  A single question assesses participants' ability to use smartphone apps on a scale of 0 to 100, with higher scores indicating greater ability to use apps on the smartphone. We hypothesize that this variable could moderate the outcome effects.
self-developed question regarding the attitude towards online interventions | baseline measurement only (week 0) before intervention starts
  To assess a person's attitude toward online circumvention, a question is asked that is rated on a scale of 0 ("not helpful at all") to 100 ("extremely helpful"), with higher scores indicating higher positive expectations. We hypothesize that this variable could moderate the outcome effects.
Client Satisfaction Questionnaire (CSQ) | Only post measurement (week 12)
  Treatment satisfaction will be measured by using the Client Satisfaction Questionnaire (CSQ), which we adapted slightly to match the use of the app. The questionnaire consists of 8 questions rated on a scale from 1 ("not at all") to 4 ("definitely yes").
Self-developed questionnaire on negative effects of treatment | Only post measurement (week 12)
  Drawing on the results of Boettcher et al., we developed a brief (7-item) scale with items covering the negative side effects that were considered most relevant by a group of experts. The items are rated on a scale from 0 ("do not agree at all") to 5 ("fully agree"). Please note, that the descriptive list of possible side effects is preliminary and may be slightly revised after the pilot study. As the list contains an open item, responses to this item will be evaluated after the pilot study and inclusion of further side effects in the list is possible should they be mentioned frequently.
Clinical Global Impression (CGI) | change from baseline to week 12 (post) and to week 36 (follow-up)
  The CGI-Severity scale provides information about the current severity of social phobic symptoms which are rated on a 7-step scale from "normal" or "not ill at all" to "among the most severely ill patients" by a clinician. The CGI-Improvement scale is a 7-point scale rating the change in symptom severity from 'improved by a lot' to 'a lot worse'. The use of the CGI, as a measure for symptom-specific improvement for patients with SAD, is supported by adequate psychometric properties and its practicability.
Quick Inventory of Depressive Symptoms (QIDS-C) | change from baseline to week 12 (post) and to week 36 (follow-up)
  The Quick Inventory of Depressive Symptomatology (QIDS-C) is a 16-item rating instrument for the assessment of depressive symptoms by an independent interviewer.
Structured Clinical Interview for DSM 5 SCID-V-CV | change from baseline to week 12 (post) and to week 36 (follow-up)
  Structured interview providing a formal diagnosis. Psychometric properties showed good reliability and specificity.
Modified version of the Social Phobia Weekly Summary Scale (SPWSS) | weekly questionnaire from baseline to week 12 (post), as well as assessments at baseline, 6 weeks (mid), 12 weeks (post), and 36 weeks (follow-up)
  Social anxiety and social approach behavior will be measured using a modified version of the Social Phobia Weekly Summary Scale (SPWSS). The individual points are rated on a scale from 0 to 100, with higher values indicating a higher rating of the respective item.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Stangier, Professor, Principal Investigator — Goethe University Frankfurt; Jürgen Hoyer, Professor, Principal Investigator — Technische Universitaet Dresden
Locations (2):
- Germany (2):
  - Technische Universitaet Dresden, Dresden
  - Goethe Universitaet Frankfurt, Frankfurt

IPD SHARING:
Plan to Share IPD: Yes
The data used in this study is available from the corresponding authors upon reasonable request.